CLINICAL TRIAL: NCT06570707
Title: Cluster-Randomized Controlled Trial (RCT) to Evaluate the Impact of a School-based Fruit and Vegetable Co-op on Cardiometabolic Health of Children and Parents in a Persistent Poverty Area
Brief Title: Evaluating the Impact of a School-based Fruit and Vegetable Co-op on Cardiometabolic Child and Parents Health in a Persistent Poverty Area
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shreela V Sharma, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0282; 5U54CA280804-02 (NIH)
Record Dates: First submitted 2024-07-31; First posted 2024-08-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Child Obesity; Cardiometabolic Health
Keywords: Brighter Bites
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brighter Bites (Experimental): This group will receive the Brighter Bites intervention throughout the study implementation. The intervention includes fruit and vegetable distributions of ~20lbs. for teachers and families, healthy recipe tastings, and nutrition education.
  Interventions: Other: Brighter Bites
- Control group (No Intervention): This delayed intervention group will receive the Brighter Bites intervention after concluding their participation in the study.

INTERVENTIONS:
Other: Brighter Bites — Families will receive a distribution of fresh fruits and vegetables (FV) (~20lbs., 50 servings/family/distribution) for ~16 weeks during the school year using primarily donated produce from local food banks. Nutrition education will be implemented for children using the evidence-based Coordinated Approach to Child Health (CATCH) program and for parents using bilingual nutrition handbooks and fun food experiences such as healthy FV recipe tastings for families during produce pick-up time will be conducted.
  Arms: Brighter Bites

SUMMARY:
The purpose of this study is to examine the effects of the (Brighter Bites (BB) intervention compared to a wait-list control group 9 months after the intervention on changes in primary child outcomes (HbA1c, and vegetable intake), on changes in secondary outcomes (household food security status, parent and child dietary behaviors, and home access/availability of fruits and vegetables (FV)), and the mediational influence of changes in food security status, parent outcomes, and home environment measures on changes in child outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of the (Brighter Bites (BB) intervention compared to wait-list control at post intervention on changes in primary child outcomes (HbA1c, and vegetable intake), to examine the effects of the BB intervention compared to wait-list control at 9-month post intervention on changes in secondary outcomes (household food security status, parent and child dietary behaviors, and home access/availability of fruits and vegetables (FV)),to examine the mediational influence of changes in food security status, parent outcomes, and home environment measures on changes in child outcomes at 9-month post-intervention, using within-subject analyses, examine and compare the long-term and dose-response effects of the BB intervention strategies on diet, adiposity, and metabolic outcomes at 21-month follow-up in the children and to explore the moderating effects of social and environmental variables on program effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* enrollment of 100 1st, 2nd, and 3rd grade students
* high proportion of children participating in the free and reduced lunch (FRL) program (>70%)
* willingness to implement a coordinated school health (CSH) program

Exclusion Criteria:

* Prior participation in BB in the previous school year
* children or parents identified as special needs per school; or having any physical, cognitive, or psychological disability that would prevent participation in evaluation measures

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in level of child Glycosylated hemoglobin (HbA1c) | baseline, post intervention (9 months after baseline)
  We will utilize the portable HbA1c analyzers (DCA Vantage analyzer) to assess HbA1c, during biometric events.
Change in amount of child vegetable intake as assessed by the VEGGIE METER® | baseline, post intervention (9 months after baseline)
  The VEGGIE METER® is used to obtain a child's quantitative metric of skin carotenoids, a proxy measure of FV intake for children. The VEGGIE METER® measures skin carotenoids as an indicator of FV intake. Higher number of carotenoid levels indicate more FV intake.

SECONDARY OUTCOMES:
Change in household food security status as assessed by a parent survey | baseline, post intervention (9 months after baseline)
  Household Food Insecurity will be measured using 2-item Hunger Vital Sign food security survey and 4-items adapted from the Center for Nutrition and Health Impact, for a total of 6-items.
  The items are scored from 0 (if the participant selects "Always") to 4 (if the participant selects "Never") and the measure's score is the mean of the responses. The higher the participant's score, the greater degree of the household nutrition security.
Number of servings consumed by the parent as assessed by the Adapted Health of Houston Survey (HHS) on processed food/drinks 4-items, and fruit and vegetable intake 2 items. | baseline, post intervention (9 months after baseline)
  This is a 6-item questionnaire. The parent responds the number of servings they consumed during the time period. Servings are calculated based on the servings per day.
Number of servings consumed by the Child as assessed by the NIH's Eating at America's Table questionnaire (All Day) and the Dietary Screener Questionnaires | baseline, post intervention (9 months after baseline)
  This is a 6-item questionnaire. The parent responds the number of servings their child consumed during the time period. Servings are calculated based on the servings per day.
Child systolic blood pressure | baseline
  Child's systolic blood pressure will be obtained with an automatic cuff according to recommendations of the American Heart Association. This will be measure during biometric events.
Child systolic blood pressure | Post intervention (9 months after baseline)
  Child's systolic blood pressure will be obtained with an automatic cuff. This will be measure during biometric events.
Child diastolic blood pressure | baseline
  Child's diastolic blood pressure will be obtained with an automatic cuff. This will be measure during biometric events.
Child diastolic blood pressure | post intervention (9 months after baseline)
  Child's diastolic blood pressure will be obtained with an automatic cuff. This will be measure during biometric events.
Change in home access/availability of fruits and vegetables as assessed by the Nutrition security measures questionnaire | baseline, post intervention (9 months after baseline)
  Nutrition security measures assess factors associated with a household's ability to obtain foods that meet their nutritional and health needs. Household Food Insecurity will be measured using 2-item Hunger Vital Sign food security survey and 4-items adapted from the Center for Nutrition and Health Impact, for a total of 6-items.
  The items are scored from 0 (if the participant selects "Always") to 4 (if the participant selects "Never") and the measure's score is the mean of the responses. The higher the participant's score, the greater degree of the household nutrition security.

CONTACTS AND LOCATIONS:
Overall Officials: Shreela Sharma, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No